CLINICAL TRIAL: NCT04463875
Title: Real World, Open Label Prospective Experience of Supplementation With a Fixed Combination of Magnesium, Vitamin B2, Feverfew, Andrographis Paniculata and Coenzyme Q10 for Episodic Migraine Prophylaxis
Brief Title: Magnesium, Vitamin B2, Feverfew, Andrographis Paniculata and Coenzyme Q10 for Episodic Migraine Prophylaxis
Status: Completed | Type: Observational
Sponsor: Corfu Headache Clinic (Other)
Responsible Party: Principal Investigator, KONSTANTINOS SPINGOS, Dr., Corfu Headache Clinic
Other Study IDs: Corfu HC
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Migraine
Keywords: episodic migraine; supplement; Vivinor; magnesium; vitamin B2; andrographis paniculata; coenzyme Q10
MeSH Terms: conditions — Migraine Disorders | interventions — Magnesium; Riboflavin; feverfew extract; Andrographis paniculata extract; coenzyme Q10

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: magnesium, vitamin B2, feverfew, andrographis paniculata and coenzyme Q10 — Supplementation per os
  Other Names: Vivinor

SUMMARY:
To investigate efficacy and safety of a supplementation with a fixed combination of magnesium, vitamin B2, feverfew, andrographis paniculata and coenzyme Q10 (Vivinor®) in episodic migraine prevention, by an observational, prospective real-world study in 113 Greek patients with episodic migraine that were prospectively followed-up for three months. The primary endpoint was the change in monthly migraine days between baseline period (BL)and the third month of treatment (T3).

DETAILED DESCRIPTION:
To investigate efficacy and safety of a supplementation with a fixed combination of magnesium, vitamin B2, feverfew, andrographis paniculata and coenzyme Q10 (Vivinor®) in episodic migraine prevention.

An observational, prospective real-world study. After a one-month baseline period, Vivinor® was introduced in 113 Greek patients with episodic migraine that were prospectively followed-up for three months. The primary endpoint was the change in monthly migraine days between baseline period (BL)and the third month of treatment (T3). Secondary endpoints included changes in mean intensity of migraine and in days with use of acute migraine medications. Changes in scores of Migraine Disability Assessment questionnaire (MIDAS), Headache Impact Test-6 (HIT-6), Migraine Therapy Assessment questionnaire (MTAQ), MSQ-QOL (Migraine-Specific Quality of life questionnaire), HADS (Hospital Anxiety and Depression Scale) were also evaluated. Those with ≥50% reduction in monthly migraine days during T3 compared to BL were considered Vivinor®-responders.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of episodic migraine with or without aura for more than one year prior to study entry
* evidence of 4-14 migraine days per month during the last trimester prior to screening
* participants may had been either treatment- naive or not suitable for or had failed previous migraine pharmacological prophylactic treatments
* were able to fully understand protocol and study information provided by the investigators.
* enrolled patients should take no other preventive treatment or use any other migraine prophylactic method during the three months before entering the study and throughout the study period.

Exclusion Criteria:

* older than 50 years of age at migraine onset
* evidence of MOH
* pregnant or nursing females
* history of tension-type, cluster or hemiplegic headache
* history of severe anaphylactic reactions to any of the intervention's ingredients
* evidence of severe systemic diseases
* history or evidence of major psychiatric disorder.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: adult patients with a documented history of episodic migraine with or without aura for more than the 12 months prior to screening, according to the criteria of the International Classification of Headaches Disorders-III (IHS, 2013)
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in monthly migraine days | 3 months
  Change in monthly migraine days between baseline period (BL) and the third month of treatment (T3)

SECONDARY OUTCOMES:
Mean intensity of migraine | 3 months
  Changes in mean intensity of migraine between baseline period (BL) and the third month of treatment (T3)
days with use of acute migraine medications | 3 months
  Changes in days with use of acute migraine medications between baseline period (BL) and the third month of treatment (T3)
Migraine Disability Assessment questionnaire (MIDAS) | 3 months
  Changes in scores of Migraine Disability Assessment questionnaire (MIDAS) during T3
Headache Impact Test-6 (HIT-6) | 3 months
  Changes in Headache Impact Test-6 (HIT-6) during T3
Migraine Therapy Assessment questionnaire (MTAQ) | 3 months
  Changes in Migraine Therapy Assessment questionnaire (MTAQ) during T3

OTHER OUTCOMES:
Migraine responders | 3 months
  Those with ≥50% reduction in monthly migraine days during T3 compared to BL were considered Vivinor®-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Michail, MD, MSc, PhD, Principal Investigator — Mediterraneo Hospital, Glyfada, Greece
Locations (1):
- Corfu HC, Corfu, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holland S, Silberstein SD, Freitag F, Dodick DW, Argoff C, Ashman E; Quality Standards Subcommittee of the American Academy of Neurology and the American Headache Society. Evidence-based guideline update: NSAIDs and other complementary treatments for episodic migraine prevention in adults: report of the Quality Standards Subcommittee of the American Academy of Neurology and the American Headache Society. Neurology. 2012 Apr 24;78(17):1346-53. doi: 10.1212/WNL.0b013e3182535d0c. PMID 22529203